CLINICAL TRIAL: NCT02138747
Title: A Prospective, Double-Blind, Randomized, Two-Period Crossover, Multi-Center Study to Evaluate the Tolerability and Patient Preference Between Myrbetriq® and Detrol® LA in Subjects With Overactive Bladder (OAB)
Brief Title: A Study to Evaluate Tolerability and Participants Preference Between Mirabegron and Tolterodine Extended Release (ER) in Participants With Overactive Bladder (OAB)
Acronym: PREFER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 178-MA-1001
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Overactive Bladder (OAB)
Keywords: Overactive bladder (OAB); tolterodine ER; mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AB: Mirabegron/Tolterodine ER (Experimental): In the treatment sequence AB participants received 25 mg of mirabegron (Myrbetriq) oral controlled absorption system (OCAS) modified-release tablets and 4 mg of placebo-to-match (PTM) tolterodine ER (Detrol LA) orally once a day during period 1. In the period 2, participants received 4 mg of tolterodine ER and 25 mg of PTM mirabegron orally once a day. Four weeks after the start of each 8-week treatment period, 25 mg of mirabegron or mirabegron PTM was increased to 50 mg for the remainder of the treatment period.
  Interventions: Drug: Mirabegron; Drug: Tolterodine ER
- BA: Tolterodine ER /Mirabegron (Experimental): In the treatment sequence BA participants received 4 mg of tolterodine ER and 25 mg of PTM mirabegron (OCAS) modified-release tablets orally once a day during period 1. In the period 2, participants received 25 mg of mirabegron and 4 mg of PTM tolterodine ER orally once a day. Four weeks after the start of each 8-week treatment period, 25 mg of mirabegron or mirabegron PTM was increased to 50 mg for the remainder of the treatment period.
  Interventions: Drug: Mirabegron; Drug: Tolterodine ER
- AA: Mirabegron/Mirabegron (Experimental): In treatment sequence AA participants received 25 mg of mirabegron and PTM tolterodine ER 4 mg capsules during period 1 and 2 orally once a day. Four weeks after the start of each 8-week treatment period, 25 mg of mirabegron was increased to 50 mg for the remainder of the treatment period.
  Interventions: Drug: Mirabegron
- BB: Tolterodine ER /Tolterodine ER (Experimental): Participants received 4 mg of tolterodine ER and PTM mirabegron 25 mg OCAS modified-release tablets orally once a day during period 1 and period 2.
  Interventions: Drug: Tolterodine ER

INTERVENTIONS:
Drug: Mirabegron — Oral
  Other Names: Myrbetriq; YM178
  Arms: AA: Mirabegron/Mirabegron; AB: Mirabegron/Tolterodine ER; BA: Tolterodine ER /Mirabegron
Drug: Tolterodine ER — Oral
  Other Names: Detrol LA
  Arms: AB: Mirabegron/Tolterodine ER; BA: Tolterodine ER /Mirabegron; BB: Tolterodine ER /Tolterodine ER

SUMMARY:
The purpose of this study was to assess tolerability of mirabegron compared to tolterodine ER in the treatment of participants with symptoms of Overactive Bladder (OAB) as well as the impact of treatment on micturition frequency and incontinence episodes.

DETAILED DESCRIPTION:
The study consisted of two double-blind treatment periods with a wash-out period in between.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to complete the micturition diary and questionnaires correctly.
* Participant has symptoms of OAB (urinary frequency and urgency with or without incontinence) for greater than or equal to 3 months prior to Screening.
* Participant must be treatment-naïve to pharmaceutical agents for OAB.
* Female participant must not donate ova starting at Screening and throughout the study period, and for 30 days after the final study drug administration.
* Male participant must not donate sperm starting at Screening and throughout the study period and for at least 30 days after final study drug administration.
* Participant agrees not to participate in another interventional study from the time of screening until the final study visit.
* Inclusion Criteria assessed at Visit 2 (Week 0) based on the 3-day micturition diary:

  * Participant continues to meet all inclusion criteria of Visit 1.
  * Participant must experience at least 3 episodes of urgency (grade 3 or 4) during the 3 day micturition diary.
  * Participant must experience an average of greater than or equal to 8 micturitions/day on the 3 day micturition diary

Exclusion Criteria:

* Female participant who is lactating or is intending to breastfeed during the study period and for 30 days after the final study visit.
* The participant has clinically significant bladder outlet obstruction (BOO) posing a risk of urinary retention.
* Participant has significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor.
* Participant has evidence of Urinary Tract Infection (UTI) (urine culture greater than 100,000 cfu/mL) as assessed at Screening (Visit 1). The participant can be rescreened after successful treatment of the UTI (confirmed by a laboratory result of negative urine culture).
* Participant has a neurological cause for detrusor overactivity (e.g., neurogenic bladder, diabetic neuropathy or systemic or central neurological disease such as multiple sclerosis and Parkinson's disease).
* Participant has an indwelling catheter or practices intermittent self-catheterization.
* Participant has a chronic inflammatory condition such as interstitial cystitis, bladder stones, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs (i.e., within the confines of the pelvis including the bladder and rectum in both sexes and the uterus, ovaries, and fallopian tubes in females); or of the lower gastrointestinal tract.
* Participant has uncontrolled narrow angle glaucoma, urinary or gastric retention, severe colitis ulcerosa, toxic megacolon, myasthenia gravis, polio or any other medical condition which makes the use of anticholinergics contraindicated.
* Participant has received intravesical injection in the past 12 months with botulinum toxin, resiniferatoxin, or capsaicin.
* Participant has received invasive treatment including electro-stimulation therapy.
* Participant is receiving a bladder training program or pelvic floor exercises which started or has changed less than 30 days prior to Screening.
* Participant has hepatic impairment defined as Child-Pugh Class A, B or C.
* Participant has severe renal impairment defined as creatinine clearance less than 30 mL/min. A participant with End Stage Renal Disease or undergoing dialysis is also not a candidate for the study.
* Participant has severe uncontrolled hypertension, which is defined as a sitting systolic blood pressure greater than or equal 180 mmHg and/or diastolic blood pressure greater than or equal 110 mmHg.
* Participant has evidence of QT prolongation on electrocardiogram (ECG) defined as QTcF greater than 450 msec for males, QTcF greater than 470 msec for females or a known history of QT prolongation.
* Participant has a serum creatinine greater than 150 µmol/L, or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2x upper limit of normal (ULN), or γ-GT greater than 3x ULN and considered clinically significant.
* Participant has a hypersensitivity to any components of Myrbetriq (mirabegron), other β-AR agonists, tolterodine or other antimuscarinic agents, or any of the inactive ingredients.
* Participant has been treated with an experimental device within 30 days or received an investigational agent within 30 days prior to Screening.
* Participant has a concurrent malignancy or history of any malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Participant with current history of alcohol and/or drug abuse.
* Participant is involved in the conduct of the study as an employee of the Astellas group, third party associated with the study, or the study site team.
* Exclusion Criteria assessed at Visit 2 (Week 0):

  * Participant fulfills any exclusion criteria at Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2015-10-29 (Actual); Study Completion 2015-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Scientific & Medical Affairs, Inc.
Locations (30):
- United States (22):
  - Site US10002 Urology Centers of Alabama, Homewood, Alabama
  - Site US10004 Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Site US10001 Urological Associates of Southern Arizona, Tucson, Arizona
  - Site US10003 Genesis Research, San Diego, California
  - Site US10010 Skyline Urology, Sherman Oaks, California
  - Site US10028 Clinical Research Consulting, Milford, Connecticut
  - Site US10024 Coastal Connecticut Research, LLC, New London, Connecticut
  - Site US10033 Eastern Research, Hialeah, Florida
  - Site US10023 Advanced Clinical Research of Miami, Miami, Florida
  - Site US10007 Pinellas Urology, Inc, St. Petersburg, Florida
  - Site US10022 Palm Beach Research Center, West Palm Beach, Florida
  - Site US10008 The Iowa Clinic PC, Urology, West Des Moines, Iowa
  - Site US10014 Mid Atlantic Clinical Research, Greenbelt, Maryland
  - Site US10005 Boston Clinical Trials, Boston, Massachusetts
  - Site US10021 AccuMed Research Associates, Garden City, New York
  - Site US10013 Advanced Urology Centers of New York, Plainview, New York
  - Site US10020 Upstate Clinical Research Associates LLC, Williamsville, New York
  - Site US10017 The Jackson Clinic, Jackson, Tennessee
  - Site US10057 Practice Research Organization, Dallas, Texas
  - Site US10035 Millennium Clinical Research Center, Arlington, Virginia
  - Site US10032 Clinical Research and Consulting Center, LLC, Fairfax, Virginia
  - Site US10034 Health Research of Hampton Roads Inc, Newport News, Virginia
- Canada (8):
  - Site CA15012 Glover Medical Clinic, Langley, British Columbia
  - Site CA15008 Silverado Research, Victoria, British Columbia
  - Site CA15003 The Male/Female Health & Research Centre, Barrie, Ontario
  - Site CA15001 Jonathan Giddens Medicine Professional Corporation, Brampton, Ontario
  - Site CA15011 Scisco Clinical Research, Cornwall, Ontario
  - Site CA15002 RechercheGCP Research, Granby, Quebec
  - Site CA15007 RechercheGCP Research, Montreal, Quebec
  - Site CA15005 CHUS - Hopital Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited participants were male and female over 18 years of age with overactive bladder (OAB) symptoms and naïve to pharmacologic treatment. The study was conducted at 36 sites (8 sites in Canada and 28 sites in the US).
Pre-assignment Details: After screening, participants were randomized into 1 of 4 sequences in a 5:5:1:1 ratio (mirabegron/tolterodine extended release (ER), tolterodine ER/mirabegron, mirabegron/mirabegron or tolterodine ER/tolterodine ER. Each participant completed 2 double-blind treatment periods with a 2-week washout period between the two periods.
Period: Treatment Period 1
Arm/Group | AB: Mirabegron/Tolterodine ER | BA: Tolterodine ER /Mirabegron | AA: Mirabegron/Mirabegron | BB: Tolterodine ER /Tolterodine ER
Started | 156 | 157 | 31 | 32
Completed | 136 | 132 | 27 | 28
Not Completed | 20 | 25 | 4 | 4
Not completed — Adverse Event | 10 | 14 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 1 | 3
Not completed — Other - Miscellaneous | 2 | 4 | 0 | 0
Period: Treatment Period 2
Arm/Group | AB: Mirabegron/Tolterodine ER | BA: Tolterodine ER /Mirabegron | AA: Mirabegron/Mirabegron | BB: Tolterodine ER /Tolterodine ER
Started | 138 (Two participants who discontinued treatment in period 1 entered period 2.) | 132 | 26 (One participant completed treatment in period 1.) | 27 (One participant completed treatment in period 1.)
Completed | 121 | 125 | 24 | 24
Not Completed | 17 | 7 | 2 | 3
Not completed — Adverse Event | 6 | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 1 | 2
Not completed — Other - Miscellaneous | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Analysis Set (RAS) included all participants who were randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | AB: Mirabegron/Tolterodine ER | BA: Tolterodine ER /Mirabegron | AA: Mirabegron/Mirabegron | BB: Tolterodine ER /Tolterodine ER | Total
Number analyzed (Participants) | 156 | 157 | 31 | 32 | 376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (14.68) | 52.6 (12.65) | 59.3 (12.95) | 55.1 (14.30) | 53.7 (13.75)
Age, Customized [Number; unit: Participants]
  < 65 Years | 119 | 129 | 20 | 23 | 291
  >= 65 Years | 37 | 28 | 11 | 9 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 119 | 19 | 22 | 277
  Male | 39 | 38 | 12 | 10 | 99
Mean Number of Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: Incontinence Episodes/24 Hours] | 3.11 (4.2) | 3.29 (4.6) | 3.76 (5.17) | 3.73 (4.92) | 3.29 (4.51)
Mean Number of Urgency Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: Urgency Incontinence Episodes] | 2.82 (4.18) | 2.83 (4.25) | 3.68 (5.19) | 3.54 (4.83) | 2.96 (4.35)
Mean Number of Micturitions per 24 Hours [Mean (Standard Deviation); unit: Micturitions] | 11.24 (2.62) | 11.65 (3.68) | 12.76 (2.63) | 11.85 (2.57) | 11.59 (3.12)
Mean Number of Urgency Episodes per 24 Hours [Mean (Standard Deviation); unit: Urgency Episodes] | 5.3 (4.1) | 5.61 (4.61) | 6.23 (4.47) | 6.29 (4.55) | 5.59 (4.38)
Mean Number of Nocturia Episodes per 24 Hours [Mean (Standard Deviation); unit: Nocturia Episodes] — Number of participants with available data in treatment groups AB, BA, AA and BB are as follows; AB=138; BA=148; AA=29; BB=30.
  Nocturia Episodes | 1.63 (1.03) | 1.49 (0.95) | 2.23 (1.05) | 1.58 (1.17) | 1.62 (1.03)
Duration of OAB Symptoms (Months) [Mean (Standard Deviation); unit: Months] | 82.75 (74.89) | 83.92 (104.56) | 73.54 (83.61) | 67.54 (58.21) | 81.19 (87.92)
Incontinence at Baseline of Period 1 [Number; unit: Participants] — Wet: at least 1 incontinence episode at baseline of period 1. Dry: 0 incontinence episodes at baseline of period 1.
  Participants
    Wet | 117 | 108 | 25 | 24 | 274
    Dry | 39 | 49 | 6 | 8 | 102
Type of OAB [Number; unit: Participants]
  Urgency | 66 | 60 | 13 | 14 | 153
  Mixed | 54 | 56 | 10 | 10 | 130
  Frequency urgency without incontinence | 36 | 41 | 8 | 8 | 93
Previous Nondrug Treatment for OAB [Number; unit: Participants]
  Yes | 6 | 6 | 1 | 3 | 16
  No | 150 | 151 | 30 | 29 | 360

OUTCOME MEASURES:

1. Primary Outcome: Participants Tolerability Assessed by the Medication Tolerability Scale of the Overactive Bladder-Satisfaction (OAB-S) Questionnaire at the End of Treatment (EOT)
Description: The medication tolerability scale measured the level of bothersomeness related to the occurrence of a side effect that was known to be related to the approved OAB medication (i.e., constipation, dry mouth, drowsiness, headache, nausea and blurred vision). The OAB medication tolerability score was calculated as a sum of the responses and converted to a scale from 0 to 100, where higher score indicates better perceived OAB medication tolerability (less bother from side-effects).
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: The Full Analysis Set (FAS) comprised of all randomized participants who received at least 1 dose of double blind study drug and had filled out OAB-S tolerability scale at least once for a postbaseline visit. Last observation carried forward imputation (LOCF) was utilized.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Groups:
- Mirabegron: Participants received 25 mg of mirabegron oral controlled absorption system (OCAS) modified-release tablets orally once a day for 8 weeks in treatment periods 1 and/or 2. Four weeks after the start of each 8-week treatment period, 25 mg of mirabegron was increased to 50 mg for the remainder of the treatment period.
- Tolterodine ER: Participants received 4 mg of tolterodine ER capsules orally once a day for 8 weeks in treatment periods 1 and/or 2.
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 341 | 336
Units on a Scale | 86.29 (1.418) | 83.40 (1.423)
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine ER; Tolerability score was analyzed using the ANOVA model (Model #1), with sequence group, study period, period-by-sequence interaction, gender and treatment group as factors, and subject-within-sequence as a random term. p-value based on the ANOVA model. Difference used mirabegron as the reference (difference =tolterodine ER -mirabegron). A negative difference indicates better reported tolerability with mirabegron than with tolterodine ER; Test type: Superiority or Other; p = 0.004, ANOVA — p-value based on the ANOVA model; LS Mean Difference = -2.89, 95% CI 2-sided [-4.86 to -0.93], Standard Error of Mean 0.997

2. Secondary Outcome: Participants Preference Based on a 5-Point Scale at the End of Period 2 in Participants Who Completed at Least 14 Days of Study Drug in Both Study Treatment Periods.
Description: Participants were asked to choose which treatment period they preferred and the degree of preference. Preference was assessed on a 5-point scale assessed at the end of period 2 ("strong preference for period 1," "mild preference for period 1," "no preference," "mild preference for period 2," "strong preference for period 2"). Participants who selected either a "mild preference" or "strong preference" were considered as having a preference for a specific study drug and participants who selected "no preference" were considered as having no preference for one study drug over the other study drug."
Time Frame: Week 18 (End of Period 2)
Population: Full Analysis Set (FAS-PNP [Preference/No Preference]) consisted of all randomized participant who took at least 14 days of double-blind study drug in each treatment period and had filled out the patient preference form.
Measure: Number; unit: Percentage of participants
Arm/Group | AB: Mirabegron/Tolterodine ER | BA: Tolterodine ER /Mirabegron | AA: Mirabegron/Mirabegron | BB: Tolterodine ER /Tolterodine ER
Number analyzed (Participants) | 127 | 125 | 25 | 26
Percentage of participants
  Preference for Period 1 | 29.9 | 34.4 | 36.0 | 23.1
  Preference for Period 2 | 37.8 | 37.6 | 36.0 | 50.0
  No Preference | 32.3 | 28.0 | 28.0 | 26.9
  Total With Preference | 67.7 | 72.0 | 72.0 | 73.1
Statistical Analysis 1: Comparison: AB: Mirabegron/Tolterodine ER vs BA: Tolterodine ER /Mirabegron; Participants who selected Mirabegron or Tolterodine ER were included in the denominator and participants with No Preference were excluded. Comparison was between Mirabegron vs Tolterodine ER; Test type: Superiority or Other; p = 0.77, Mainland-Gart — P value was obtained using Mainland-Gart test to compare the proportion of preference for each treatment group. The denominator excluded patients with No Preference

3. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: Impact on Daily Living With OAB.
Description: Impact on daily living with the OAB was scored from 0 to 100, with higher scores indicating greater satisfaction with ability to perform daily activities.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: Full Analysis Set (FAS) consisted of all randomized patients who received at least 1 dose of double blind study drug and had filled out OAB-S tolerability scale at least once for a post baseline visit. Last observation carried forward imputation (LOCF) was utilized.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Units on a Scale | 72.98 (1.419) | 71.92 (1.521)

4. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: OAB Control
Description: OAB control was scored from 0 to 100, with higher scores indicating better OAB control.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: Full Analysis Set (FAS) consisted of all randomized patients who received at least 1 dose of double blind study drug and had filled out OAB-S tolerability scale at least once for a postbaseline visit. Last observation carried forward imputation (LOCF) was utilized.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Units on a Scale | 64.49 (1.205) | 63.38 (1.266)

5. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: Satisfaction With OAB Control
Description: Satisfaction with OAB control was scored from 0 to 100 with higher scores indicating greater satisfaction with OAB control.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Units on a Scale | 69.17 (1.491) | 68.31 (1.524)

6. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: Overall Assessment of Participant's Fulfillment of OAB Medication Expectations
Description: The final item score for overall assessment of patient's fulfillment of OAB medication expectations ranged from 1 to 5, with higher scores indicating better fulfillment of OAB medication expectations.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Units on a Scale | 3.10 (0.072) | 3.08 (0.073)

7. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: Overall Assessment of Interruption of Day-to-Day Life Due to OAB
Description: Overall assessment of interruption of day-to-day life due to OAB was assessed on a scale from 1 to 5, with higher scores indicating less interruption of day-to-day life due to OAB symptoms.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Unit on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Unit on a Scale | 3.00 (0.068) | 3.02 (0.067)

8. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: Overall Satisfaction With OAB Medication
Description: Overall satisfaction with OAB medication was assessed on a scale of 1 to 5, with higher scores indicating greater satisfaction with current OAB medication.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Units on a Scale | 3.70 (0.071) | 3.66 (0.074)

9. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: Overall Assessment of Willingness to Continue OAB Medication
Description: Overall assessment of willingness to continue OAB medication, was assessed on a scale from 1 to 5, with higher scores indicating greater desire to continue with current OAB medication.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Units on a Scale | 3.69 (0.071) | 3.69 (0.071)

10. Secondary Outcome: Scale of the OAB-S Questionnaire at the End of Treatment Period: Overall Assessment of Improvement in Day-to-Day Life Due to OAB Medication
Description: Overall assessment of improvement in day-to-day life due to OAB medication was assessed on a scale from 1 to 5, with higher scores indicating greater improvement in day-to-day life due to current OAB medication.
Time Frame: Week 8 (End of Period 1) and Week 18 (End of Period 2)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 336 | 330
Units on a Scale | 3.43 (0.079) | 3.46 (0.078)

11. Secondary Outcome: Change From Baseline to End of Treatment (EOT) in Mean Number of Incontinence Episodes Per 24 Hours
Time Frame: Baseline and EOT (Period 1-Week 8 and Period 2- Week 18)
Population: Full Analysis Set Incontinence (FAS I) consisted of all participants in the FAS who had at least 1 incontinence episode in the baseline 3-day micturition diary and at least 1 postbaseline diary during period 1.Last observation carried forward imputation (LOCF) was utilized.
Measure: Least Squares Mean (Standard Error); unit: Incontinence Episodes
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 243 | 233
Incontinence Episodes | -1.51 (0.194) | -1.46 (0.194)
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine ER; Adjusted difference vs mirabegron where difference used mirabegron as the reference (difference = tolterodine ER - mirabegron); Test type: Superiority or Other; p = 0.971, ANCOVA — Adjusted P value was generated from the ANCOVA model for the period-by-treatment interaction; LS Mean Difference = 0.05, 95% CI 2-sided [-0.39 to 0.49], Standard Error of Mean 0.224

12. Secondary Outcome: Change From Baseline to End of Treatment (EOT) in Number of Micturitions Per 24 Hours
Time Frame: Baseline and EOT (Period 1-Week 8 and Period 2- Week 18)
Population: Full Analysis Set (FAS) consisted of all randomized participants who received at least 1 dose of double blind study drug and had filled out OAB-S tolerability scale at least once for a post baseline visit.
  Last observation carried forward imputation (LOCF) was utilized.
Measure: Least Squares Mean (Standard Error); unit: Micturitions
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 331 | 327
Micturitions | -2.06 (0.194) | -1.95 (0.195)
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine ER; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.211, ANCOVA — Adjusted P value was generated from the ANCOVA model for the period-by-treatment interaction; LS Mean Difference = 0.11, 95% CI 2-sided [-0.28 to 0.50], Standard Error of Mean 0.199

13. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety was assessed by evaluation of treatment-emergent adverse events (TEAEs; frequency, severity, seriousness and relationship to study drug), AEs of special interest, vital signs (SBP, DBP, body temperature and pulse rate) and laboratory tests (liver function tests [LFTs]). Treatment-Emergent Adverse Event (TEAEs) were defined as any adverse event starting or worsening in the period from first dose of double-blind study drug until 15 days after last dose of double-blind study drug.
Time Frame: Baseline to EOT (Week 18) and follow up (Week 20)
Population: Safety Analysis Set consisted of all participants who received at least 1 dose of double-blind study drug (SAF).
Measure: Number; unit: Participants
Arm/Group | Mirabegron | Tolterodine ER
Number analyzed (Participants) | 319 | 325
Participants
  Adverse Events (AEs) | 150 | 168
  Drug-related (AEs) | 89 | 111
  Deaths | 0 | 0
  Serious Adverse Event (SAE) | 3 | 8
  Drug-related SAEs | 2 | 0
  AEs Leading to Permanent Discontinuation of Drug | 15 | 20
  Drug-related AEs Leading to Permanent Discontinuat | 12 | 12
  SAEs Leading to Permanent Discontinuation | 0 | 5
  Drug-related SAEs Leading to Permanent Discontinu | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to End of Treatment (Week 18) and follow up 2 weeks after (Week 20)
Description: Treatment-emergent adverse events are defined as any adverse event starting or worsening in the period from first dose double-blind study drug until 15 days after last dose of double-blind study drug. If a participant reported TEAE for the same treatment in two different periods (sequences AA/BB), then that participant was counted once.
Arm/Group | Mirabegron | Tolterodine ER
Serious Adverse Events (participants affected / at risk) | 3/319 | 8/325
Other Adverse Events (participants affected / at risk) | 55/319 | 79/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron (N=319) | Tolterodine ER (N=325)
Atrial fibrillation (Cardiac disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron (N=319) | Tolterodine ER (N=325)
Dry mouth (Gastrointestinal disorders) | 29 | 53 — If a patient reported a TEAE for the same treatment in 2 different periods, then that patient was counted once.
Constipation (Gastrointestinal disorders) | 18 | 20 — If a patient reported a TEAE for the same treatment in 2 different periods, then that patient was counted once.
Headache (Nervous system disorders) | 18 | 19 — If a patient reported a TEAE for the same treatment in 2 different periods, then that patient was counted once.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after primary publication of the multi-site data. Sponsor must receive a site's manuscript at least 45 days prior to planned submission to ensure that no confidential information of Sponsor is included in the document. In addition if requested by sponsor any publication or presentation shall be delayed for a period not to exceed 60 days.